CLINICAL TRIAL: NCT04391855
Title: Effect of Wound Infiltration With Tramadol, Dexmedetomidine, or Magnesium Sulfate as Adjuncts to the Local Anesthetic on Pain Relief After Spine Surgery
Brief Title: Wound Infiltration With Tramadol, Dexmedetomidine, or Magnesium Plus Ropivacaine for Pain Relief After Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Georgia Tsaousi, Associate Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SpinInf
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Analgesia; Pain, Postoperative; Spinal Stenosis; Spinal Disease
Keywords: analgesia; pain score; tramadol; dexmedetomidine; magnesium; opioid consumption; spine surgery
MeSH Terms: conditions — Agnosia; Pain, Postoperative; Spinal Stenosis; Spinal Diseases | interventions — Tramadol; Ropivacaine; Dexmedetomidine; Magnesium; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tramadol with ropivacaine (Experimental): Tramadol 2mg/kg with ropivacaine (10mg/ml) 100mg for wound infiltration
  Interventions: Drug: Tramadol with ropivacaine
- Dexmedetomidine with ropivacaine (Experimental): Dexmedetomidine 1μg/kg with ropivacaine (10mg/ml) 100mg for wound infiltration
  Interventions: Drug: Dexmedetomidine with ropivacaine
- Magnesium with ropivacaine (Experimental): Magnesium sulfate 10 mg/kg with ropivacaine (10mg/ml) 100mg for wound infiltration
  Interventions: Drug: Magnesium with ropivacaine
- Placebo with ropivacaine (Placebo Comparator): Ropivacaine (10mg/ml) 100mg with 5ml isotonic saline for wound infiltration
  Interventions: Drug: Ropivacaine plus normal saline

INTERVENTIONS:
Drug: Tramadol with ropivacaine — A solution of tramadol 2mg/kg with ropivacaine hydrochloride (10mg/ml) 100mg mixture making up a total volume of 15ml will be infiltrated in the surgical trauma area before closure.
  Other Names: TR
  Arms: Tramadol with ropivacaine
Drug: Dexmedetomidine with ropivacaine — A solution of dexmedetomidine 1μg/kg with ropivacaine hydrochloride (10mg/ml) 100mg mixture making up a total volume of 15ml will be infiltrated in the surgical trauma area before closure.
  Other Names: DR
  Arms: Dexmedetomidine with ropivacaine
Drug: Magnesium with ropivacaine — A solution of magnesium 10 mg/kg with ropivacaine hydrochloride (10mg/ml) 100mg mixture making up a total volume of 15ml will be infiltrated in the surgical trauma area before closure.
  Other Names: MR
  Arms: Magnesium with ropivacaine
Drug: Ropivacaine plus normal saline — A solution of ropivacaine hydrochloride (10mg/ml) 100mg with 5ml of isotonic saline 0.9% mixture making up a total volume of 15ml will be infiltrated in the surgical trauma area before closure.
  Other Names: R
  Arms: Placebo with ropivacaine

SUMMARY:
The rationale for multimodal analgesia is to achieve additive or synergistic analgesic properties while decreasing the incidence of side effects by reducing the dose of each agent. Nociceptive stimuli are known to activate the release of the excitatory amino acid glutamate in the dorsal horn of the spinal cord. The resultant activation of NMDA receptors causes calcium entry into the cell and triggers central sensitization. This mechanism is involved in the perception of pain and mainly accounts for its persistence during the postoperative period.

Peri-incisional injection of local anesthetics is an effective method for pain relief after many surgical procedures, as it can reduce postoperative analgesic consumption. Ropivacaine is a propyl analog of bupivacaine with a longer duration of action with a much safer cardiotoxicity profile than bupivacaine. Thus, a combination of local anesthetic with other analgesic factors, such as opioids, dexmedetomidine, clonidine, ketamine, magnesium sulfate, dexamethasone is suggested for a better analgesic outcome.

Dexmedetomidine, a highly selective a2-adrenergic receptor agonist, has been the focus of interest for its broad spectrum (sedative, analgesic, and anesthetic sparing) properties, making it a useful and safe adjunct in many clinical applications. The intravenous, intramuscular, intrathecal, epidural, and perineural use of this agent enhances analgesic effects.

Tramadol hydrochloride is a synthetic analog of codeine that acts on both opioid (weak m receptor agonist) and nonopioid receptors (inhibits the reuptake of noradrenaline and serotonin as well as release stored serotonin from nerve endings) which play a crucial role in pain inhibition pathway. It also blocks nerve conduction which imparts its local anesthetics like action on peripheral nerves.

It was reported that NMDA antagonists could prolong the analgesic effect of bupivacaine to even a week, as well as inhibit hyperalgesia. Magnesium sulfate (MGS) is a non-competitive antagonist of N-methyl, D-aspartate (NMDA) receptors with an analgesic effect and is essential for the release of acetylcholine from the presynaptic terminals and, similar to calcium channel blockers (CCB), can prevent the entry of calcium into the cell.

Aim of the study is to evaluate and compare the postoperative analgesic efficacy of tramadol, dexmedetomidine, and magnesium when added to ropivacaine as an adjuvant for wound infiltration following spine surgery.

DETAILED DESCRIPTION:
Each participant will receive standard monitoring (ECG, SpO2, capnography, SBP, oesophageal temperature) and intravenous access will be established. A standard anesthesia protocol will be applied involving propofol 2mg/kg (iv) and remifentanil in TCI (target-controlled infusion). Cis-atracurium 0.2 mg/kg (iv) will be given to facilitate endotracheal intubation. Anesthesia will be maintained with desflurane in a 50% air/O2 mixture A standard anesthesia protocol will be applied involving propofol 2mg/kg (iv) and remifentanil in TCI (target-controlled infusion). Cis-atracurium 0.2 mg/kg (iv) will be given to facilitate endotracheal intubation. Anesthesia will be maintained with air to oxygen mixture of 50%, and desflurane adjusted to achieve a target BIS between 40 and 50. Remifentanil target level will be titrated according to analgesic demands defined by a > 20% change of heart rate or blood pressure compared with baseline. The duration of both anesthesia and surgical procedure will be registered. Furthermore, the level of sedation upon anesthesia emergence will be recorded using the Ramsey sedation scale.

Postoperatively pain assessment will be performed by the Visual Analogue Scale (VAS) and Numerical Rating Scale (NRS) at anesthesia emergence and at 2, 4, 6, 12, 18, and 24 h after surgery conclusion. Time to first analgesic request and total analgesics consumption postoperatively (morphine equivalents) will be recorded.

Episodes of shivering, as well as episodes of nausea and vomiting (PONV) and other postoperative adverse events, will be recorded at emergence and 24 hours thereafter.

Finally, patients' global satisfaction will be assessed the second day and one month after surgery using the Quality of Recovery Scale(QoR-40). In the meantime, blood samples will be taken at the time before the surgical stimulus, 6 hours and 24 hours after wound infiltration to measure cortisol, TNF-a, and IL-6 plasma concentration.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 18 and 80 years
* ASA Physical status 1 to 3
* Elective or semi-elective one-level lumbar laminectomy or discectomy surgery
* Signed informed consent

Exclusion Criteria:

* Chronic use of opioids
* Drugs or alcohol abuse
* Neurological disorders
* Local anesthetics toxicity
* Myopathy
* Cardiac conductance disturbances
* Hepatic failure
* Renal failure
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Time to first analgesic request in minutes | 24 hours after the emergence from anesthesia
  The difference in the time frame (minutes) for analgesia request after emergence from anesthesia after wound infiltration with tramadol plus ropivacaine, tramadol plus ropivacaine, magnesium sulfate plus ropivacaine or ropivacaine plus isotonic saline 0.9%

SECONDARY OUTCOMES:
Pain intensity postoperatively | At 10 minutes after emergence from anesthesia, and 2, 4, 6, 12, 18 and 24 hours after the emergence from anesthesia
  The difference in pain intensity postoperatively assessed by Visual Analogue Scale (graded from 0 defining absence of pain to 10 meaning extreme pain) or Numerical Pain Scale (graded from 0 defining no pain to 10 the worst pain ever experienced) after wound infiltration with tramadol plus ropivacaine, tramadol plus ropivacaine, magnesium sulfate plus ropivacaine or ropivacaine plus isotonic saline 0.9%
Analgesics consumption postoperatively in morphine equivalents | 24 hours after the emergence from anesthesia
  The difference in analgesic consumption (assessed as mg of morphine equivalents) postoperatively after wound infiltration with tramadol plus ropivacaine, tramadol plus ropivacaine, magnesium sulfate plus ropivacaine or ropivacaine plus isotonic saline 0.9%
Plasma concentration of TNF-a and IL-6 | Before wound infiltration, and at 6 and 24 hours thereafter
  Levels of TNF-a and IL-6 in pg/ml will be measured from blood samples at the times before surgical stimulus, at 6 hours and 24 hours after wound infiltration, as stress-response biomarkers.
Plasma concentration of cortisol | Before wound infiltration, and at 6 and 24 hours thereafter
  Levels of cortisol (in mcg/dL) will be measured from blood samples at the times before surgical stimulus, at 6 hours and 24 hours after wound infiltration, as stress-response biomarkers.

OTHER OUTCOMES:
Patients' sedation level after emergence | At 5 minutes after emergence from anesthesia
  The level of sedation will be assessed after emergence using the Ramsey sedation scale in each participant, which ranges between 1 (anxious and restless patient) to 6 (unresponsive patient).
Postoperative adverse effects | 24 hours after the emergence from anesthesia
  The incidence of shivering, pruritus, nausea /vomiting, or any other adverse effect postoperatively after wound infiltration with tramadol plus ropivacaine, tramadol plus ropivacaine, magnesium sulfate plus ropivacaine or ropivacaine plus isotonic saline 0.9%
Quality of Recovery | At 48 hours postoperatively and one month after hospital discharge
  The quality of recovery and overall satisfaction of each participant will be assessed using the Quality of Recovery Scale (QoR-40) ranging from 0 the worst to 200 the best value.

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Tsaousi, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No